CLINICAL TRIAL: NCT01656044
Title: The Effect of Negative Pressure Therapy on Incisional Surgical Site Infections
Brief Title: Negative Pressure Therapy in Preventing Infection After Surgery in Patients With Colon, Rectal, Pancreatic, or Peritoneal Surface Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00020105; NCI-2012-00624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99212 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Colon Cancer; Pancreatic Cancer; Perioperative/Postoperative Complications; Primary Peritoneal Cavity Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Pancreatic Neoplasms; Postoperative Complications; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (SSD) (Active Comparator): Patients receive SSD over their closed laparotomy incision at the conclusion of their surgery.
  Interventions: Procedure: wound care management
- Arm II (NPT) (Experimental): Patients receive NPT dressing over their closed laparotomy incision at the conclusion of their surgery.
  Interventions: Procedure: wound care management

INTERVENTIONS:
Procedure: wound care management — Receive SSD
  Arms: Arm I (SSD)
Procedure: wound care management — Receive NPT
  Arms: Arm II (NPT)

SUMMARY:
The purpose of this research study is to evaluate if a negative-pressure dressing placed over a surgical incision can reduce the risk of developing a surgical site infection compared to a commonly-used sterile gauze incision dressing. In this study, the negative-pressure dressing will be compared to a standard post-surgical sterile gauze dressing. In this study patients will either receive a negative-pressure dressing or a standard sterile gauze dressing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether negative pressure therapy applied to closed laparotomy incisions can decrease the incidence of incisional surgical site infections in patients undergoing clean-contaminated resections for colorectal, pancreatic, and peritoneal surface malignancies compared to standard post-operative sterile gauze dressings.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive standard sterile dressing (SSD) over their closed laparotomy incision at the conclusion of their surgery.

ARM II: Patients receive negative pressure therapy (NPT) dressing over their closed laparotomy incision at the conclusion of their surgery.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Surgical resection for a colorectal, pancreatic, or peritoneal surface malignancy
* The scheduled procedure will be performed via midline laparotomy
* The planned procedure is a clean-contaminated (class II) case (includes gastric, small bowel, and colorectal resections, as well as bile or pancreatic duct transections)
* Ability to understand and the willingness to sign a written informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Emergent cases will not be included in the study
* Pregnant patients will not be included in the study as pregnancy is a relative contraindication for these types of surgical procedures
* Clean (class I), contaminated (class III) and dirty (class IV) procedures will likewise be excluded
* Patients on chronic immunosuppressive medications, including steroids, within the past three months
* Patients with a history of skin allergy to iodine or adhesive drapes
* The planned procedure involves foreign material (such as mesh or subcutaneous drains) being left in the subcutaneous space at the time of surgery (for example, a ventral hernia repair); surgical drains that are placed to drain an intraabdominal space and exit the abdominal wall remote from the incision are allowed in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2012-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Rate of incisional surgical site infection (SSI), which includes superficial incisional SSIs and deep incisional SSIs as defined by the Center of Disease Control and Prevention | 30 days
  Results will be analyzed initially using descriptive statistics. The proportion of SSI in the NPT group will be compared to the standard post-operative dressing group using a chi square test of proportions.

SECONDARY OUTCOMES:
Rates of organ/space SSIs, seromas, hematomas, incisional cellulitis, and wound opening for any reason | 30 days
The cost of NPT and SSD, as well as estimate additional costs associated with incisional SSIs in affected patients | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Perry Shen, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States